CLINICAL TRIAL: NCT04309773
Title: Double Blind, Multicentric, Randomized, Placebo-controlled Trial, Evaluating the Efficacy of 24 Month of Bezafibrate in Primary Sclerosing Cholangitis With Persistent Cholestasis Despite Ursodeoxycholic Acid Therapy
Brief Title: Efficacy of 24 Month of Bezafibrate in Primary Sclerosing Cholangitis With Persistent Cholestasis Despite Ursodeoxycholic Acid Therapy
Acronym: BEZASCLER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP180668
Record Dates: First submitted 2019-10-18; First posted 2020-03-16 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Primary Sclerosing Cholangitis; Cholestasis
Keywords: Primary sclerosing cholangitis; Persistent cholestasis; Bezafibrates; Fibrates; UDCA
MeSH Terms: conditions — Cholangitis, Sclerosing; Cholestasis | interventions — Bezafibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bezafibrate in addition to standard UDCA therapy (Experimental): Bezafibrate (400mg) in addition to standard 15-20 mg/kg/day UDCA therapy ("experimental" arm)
  Interventions: Drug: Bezafibrate (400mg) in addition to standard 15-20 mg/kg/jour UDCA therapy
- Placebo of Bezafibrate in addition to standard UDCA therapy (Placebo Comparator): Placebo of Bezafibrate in addition to standard 15-20 mg/kg/day UDCA therapy
  Interventions: Drug: Placebo of Bezafibrate in addition to standard UDCA therapy

INTERVENTIONS:
Drug: Bezafibrate (400mg) in addition to standard 15-20 mg/kg/jour UDCA therapy — Bezafibrate (400mg) in addition to standard 15-20 mg/kg/jour UDCA therapy Treatment duration : 24 months Bezafibrate/AUDC : daily oral dose
  Arms: Bezafibrate in addition to standard UDCA therapy
Drug: Placebo of Bezafibrate in addition to standard UDCA therapy — Placebo of Bezafibrate (400mg) in addition to standard 15-20 mg/kg/Day UDCA therapy Treatment duration : 24 months Placebo/AUDC : daily oral dose
  Arms: Placebo of Bezafibrate in addition to standard UDCA therapy

SUMMARY:
The objectives of this study are to evaluate the effect of bezafibrate treatment compared to placebo on efficacy and safety in patients with primary sclerosing cholangitis (PSC) and persistent cholestasis despite ursodeoxycholic acid therapy

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, evaluation of the efficacy and safety of Bezafibrate in subjects with PSC and persistent cholestasis despite ursodeoxycholic acid therapy (UADC).

Design:

* A multicentre, double-blind placebo controlled, randomised clinical trial
* 35 centers participants to the recruitment (French Network of Reference and Competence Centers for Rare Diseases: "inflammatory biliary diseases and autoimmune hepatitis" (MIVBH), including Saint-Antoine hospital, Paris as reference coordinator center)

Sample size :

104 patients, 52 in each group

Treatments groups:

1. UADC therapy (15-20 mg/kg/d) + Bezafibrate (400mg/d)
2. UDCA therapy (15-20 mg/kg/d) + placebo of bezafibrate (400mg/d)

Treatments duration :

24 months

Assessement:

Study visits at Inclusion, (M0) Randomisation and then every 3 months until M24

This is a phase III randomized, double blinded, multicenter, study.

No interim analysis is planned. Analysis will be performed at the end of the study after data review and freezing of data base according to intent to treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Males or females ≥ 18 and ≤ 75 years
* Large duct PSC verified by retrograde, operative, percutaneous or magnetic resonance cholangiography (MRC) demonstrating intrahepatic and /or extrahepatic biliary duct changes consistent with PSC
* Colonoscopy (already done or scheduled before randomization) within the last 5 years (or within 6 months if IBD is associated to PSC) with neither cancer nor allgrade dysplasia or endoscopy of the ileal reservoir (already done or scheduled before randomization) within the last 2 years in patients with ileo-anal anastomosis
* ALP ≥ 1.5 ULN at baseline
* Treatment with stable dose of UDCA (15-20 mg/kg/d) for ≥ 6 months before inclusion (rounded to the nearest unit, e.g 14.5 mg/kg/d would be 15mg/kg/d).
* Using contraceptive in childbearing women
* Affiliation to a social security system (AME excepted)
* Signed informed consent

Exclusion Criteria:

* Child-Pugh score B or C
* Ascites or digestive hemorrhage (or history of)
* Total bilirubin in the last 3 months > 50 μmole/L (3 mg/dl)
* Gilbert syndrome defined as unconjugated bilirubinemia > 12 μmol/L
* Albumin in the last 3 months < ULN (according to the laboratory reference value)
* Prothrombin index in the last 3 months < 70%
* Platelets count in the last 3 months < 100000/mm3
* ALT or AST > 5 ULN in the last 3 months
* Prior liver transplantation
* Treatment with a fibrate within the last 3 months inclusion or with a statin at inclusion
* Current active IBD defined as either current use of systemic corticosteroid therapy > 10 mg/day or budesonide > 3 mg /day or immunosuppressive drugs (cyclosporine, tacrolimus, mycophenolate mofetil, mTor inhibitors, JAK inhibitors) or a partial Mayo score > 2 in patients with ulcerative colitis (UC) or a Crohn's Disease Activity Index (CDAI) > 150 in patients with Crohn's disease (CD)
* Dose change of treatment for associated IBD ≤3 months prior to inclusion
* Current or history of colonic cancer or all-grade dysplasia described at the last colonoscopy (Patients with a history of colon cancer and treated by total colectomy without recurrence for at least 5 years are eligible)
* Any other cause of liver damage ((positive test for HBV, HCV, or HIV, excessive alcohol consumption, hemochromatosis, Wilson's disease, α1-antitrypsin deficiency, celiac disease, autoimmune hepatitis defined by the presence of at least 2 of the 3 following criteria; 1) AST or ALT > 5 ULN, 2) Positive anti smooth muscle auto antibodies or serum IgG > 1.5 ULN, 3) interface hepatitis on liver biopsy)
* Secondary causes of sclerosing cholangitis including IgG4-associated cholangitis (elevated serum IgG4 > 4 ULN)
* History of acute cholangitis in the last 3 months prior to inclusion or current acute cholangitis
* Endoscopic treatment for bile duct stenosis ≤ 3 months prior to inclusion or planned within 3 months post randomization date
* History of or established or suspected hepatobiliary carcinoma.
* Any severe comorbidity that may reduce life expectancy
* History of malignancy diagnosed or treated within 2 years (recent localized treatment of squamous or non-invasive basal skin cancers is permitted; cervical carcinoma in situ is allowed if appropriately treated prior to Screening)
* Known hypersensitivity to bezafibrate, any of the components of Befizal© or other fibrates
* Known photosensitivity or photoallergy reactions to fibrate
* Patient with congenital galactosemia, glucose malabsorption, or lactase deficiency because of presence of lactose in 400 mg SR tablets of bezafibrate and in placebo tablets
* Pregnancy (or desire for)
* Renal insufficiency (clearance < 60 ml/min or serum creatinine level > 130 μmole/L)
* Breastfeeding
* Participation in any other interventional study or in the exclusion period any other interventional study
* Autoimmune hepatitis defined by the presence of interface hepatitis documented on liver biopsy and at least 1 of the 2 following criteria: 1) AST or ALT > 5 ULN, 2) Positive anti smooth muscle auto antibodies or serum IgG > 1.5 ULN
* Results of colonoscopy not available or > 5 years (or > 6 months if IBD is associated to PSC) or with cancer or all-grade dysplasia or results of endoscopy of the ileal reservoir not available or > 2 years in patients with ileo-anal anastomosis

Randomization exclusion criteria:

* Positive test for HBV (positive HBs Ag), HCV (positive HCV RNA), or HIV (positive serology)
* Pregnancy (or desire for in the 2 next years)
* Secondary causes of sclerosing cholangitis including IgG4-associated cholangitis (elevated serum IgG4 > 4 ULN)
* Autoimmune hepatitis defined by the presence of interface hepatitis documented on liver biopsy and at least 1 of the 2 following criteria: 1) AST or ALT > 5 ULN, 2) Positive anti smooth muscle auto antibodies or serum IgG > 1.5 ULN
* Current acute cholangitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of 24-month treatment with bezafibrate (400 mg/day) versus placebo in addition to standard UDCA therapy in Primary Sclerosing Cholangitis (PSC). | At 24 months
  Proportion of patients with serum Alkaline Phosphatase < 1.5 ULN and a reduction of at least 15% from baseline at M24 and normal serum bilirubin and no increase of liver stiffness at M24 compared to baseline:

SECONDARY OUTCOMES:
Percentage of patients with clinical or biological adverse events | At 24 months
  Safety endpoint: Percentage of patients with clinical (including increased IBD activity) or biological adverse events (elevated creatinine (> 150 μmol/L) or ALT (> 5ULN) or AST (> 5ULN) or CPK (> 5ULN) during the study period.
Quality of life of PSC patients | At 12 months and 24 months
  French version of the quality of life QMCF questionnaire.
Score for pruritus | At 12 months and 24 months
  Absolute changes in the score for pruritus (measured by VAS and 5D pruritus scale) at each study visit.
Fatigue score | At 12 months and 24 months
  Absolute changes in the score for fatigue (measured by adapted PBC-40 questionnaire)
Level of liver biochemical parameters between the two groups of patient | between month 0 and month 24
  The course during the study will be studied using linear regression mixed model.
  A random effect for each patient will be considered and treatment group will be considered as fixed effects.
Occurrence of clinical events and transplant-free survival | At 24 months
  Survival rate without liver transplantation or hepatic events (ascites, variceal bleeding, encephalopathy, acute cholangitis, cholangiocarcinoma, hepatocellular carcinoma or serum total bilirubin > 100 μmol/L for at least 3 months).

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHAZOUILLERES, professor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hepatology department - Hopital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No